CLINICAL TRIAL: NCT07224451
Title: Liquid Biopsy Following Blood-Brain Barrier Disruption Using Barrier Disrupting Fields in Patients Undergoing Spine Surgery
Brief Title: Liquid Biopsy Following BBB Disruption Using Barrier Disrupting Fields in Patients Undergoing Spine Surgery
Acronym: BDF002
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Ran Harel, Director of Spine Surgery Division, Department of Neurosurgery Sheba Medical Center, Israel, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA - 25 - 2323 - RH - CTIL
Record Dates: First submitted 2025-11-03; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Spinal Tumors
Keywords: Barrier disrupting fields; pulse electrical fields; blood-brain barrier opening; blood-arachnoid barrier opening; liquid biopsy; spinal tumors
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Masking Description: The subcontractor laboratories assessing the blood and CSF samples will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- BDF are applied following anaesthesia, blood/CSF samples acquired (Experimental): Following anaesthesia a blood sample will be acquired, followed by BDF, following by additional blood samples acquisition and finally a CSF sample when opening the dura
  Interventions: Procedure: spinal surgery; Device: BDF

INTERVENTIONS:
Procedure: spinal surgery — Candidates for intradural tumor resection spinal surgery with intraoperative neuromonitoring will be enrolled in the study prior to surgery. The patient will undergo preparation for surgery according to the standard care. Once anesthetized and intubated, electrodes will be attached to the patient's head. After placing the electrodes, when the patient is under anesthesia, a blood sample will be taken prior to BDF. This sample will be used as baseline for BDF. The patient will then undergo a BDF procedure. Additional blood samples will be taken for identification of CNS biomarkers. Surgery will then proceed according to the standard of care. Once the dura is opened, a CSF sample will be taken. The surgery will continue according to the standard of care
  Other Names: Barrier disrupting fields; Acquire blood samples; Acquire CSF sample
Device: BDF — electrodes couples (voltage and ground) will be placed on the patient head and will be connected to a pulse generator. 2 electrodes couples will be activated in parallel, up to 8 electrodes couples total. EEG will be acquired after each series of pulses for a few sec.
  Other Names: pulsed electric fields

SUMMARY:
Objective: To identify new central nervous system (CNS) biomarkers to be used for blood-derived liquid biopsy once the blood-brain barrier (BBB), specifically the blood-arachnoid barrier (BAB), has been transiently disrupted by BDF in patients undergoing spine surgery.

Design: Single center (Sheba Medical Center), prospective, controlled. Phase: Feasibility study

Endpoints:

Efficacy The primary endpoint of the study is the elevation in blood concentration of CNS biomarkers following the study procedure compared to biomarkers detected in cerebrospinal fluid (CSF) of the same subject.

Safety The primary safety endpoint will be the overall incidence of BDF procedure-related AEs and SAEs, with severity graded according to CTCAE v5.0 criteria.

Study population:

The study population will include up to 20 patients undergoing spine surgery.

Study period:

24 months.

Inclusion criteria:

1. Adult subjects over the age of 18
2. Able to sign informed consent
3. Candidates for intradural tumor resection spinal surgery with intraoperative neuromonitoring.

Exclusion criteria:

1. Pacemakers, or other implanted electric medical devices
2. Pregnant or lactating females
3. Major medical, neurologic or psychiatric condition who are judged as unable to fully comply with the study
4. History of skull fractures or previous brain surgery
5. American Society of Anesthesiologists grade >2
6. Anticoagulants treatment
7. Damage to the dura resulting in CSF leak
8. Patients with seizures/epilepsy

Study procedure:

1. Candidates for intradural tumor resection spinal surgery with intraoperative neuromonitoring will be enrolled in the study prior to surgery.
2. The patient will undergo preparation for surgery according to the standard care.
3. Once anesthetized and intubated, electrodes will be attached to the patient's head.
4. After placing the electrodes, when the patient is under anesthesia, a blood sample will be taken prior to BDF. This sample will be used as baseline for BDF.
5. The patient will then undergo a BDF procedure.
6. Additional blood samples will be taken for identification of CNS biomarkers.
7. Surgery will then proceed according to the standard of care.
8. Once the dura is opened, a CSF sample will be taken, in order to compare the blood biomarkers of the specific subject with the CSF biomarkers.
9. The surgery will continue according to the standard of care.

DETAILED DESCRIPTION:
Barrier-disrupting fields (BDF), based on low pulsed electric fields, offer a non-invasive and transient method for selectively opening CNS barriers. We have previously shown that BDF can be applied for efficient delivery of systemically administered drugs into the CNS in rodents. We further demonstrated the application of BDF to enable blood-based detection of brain-derived proteins in rats and mice.

The primary endpoint of the study is the elevation in blood concentration of CNS biomarkers following the study procedure compared to biomarkers detected in CSF of the same subject. The concentration of the biomarkers is expected to be elevated in the blood after the BDF procedure. These include specific CSF proteins such as Protein S100A, S100B and prostaglandin D2 isomerase and include additional proteins identified by us in preclinical experiments in rats, and other CNS-derived molecules that were not identified in our preliminary studies.

Candidates for intradural tumor resection spinal surgery with intraoperative neuromonitoring will be enrolled in the study prior to surgery.

BDF treatment parameters are planned using a simulation package. The distributions of electric fields on the BAB are calculated using a finite elements model, to reach desired electric fields on the BAB needed for inducing BAB disruption. This is done using a simulation package, based on brain MRI after tissue segmentation. Different locations, sizes and distances between the electrodes are modeled in order to reach the optimal setup for obtaining optimal BAB disruption with no BBB disruption.

The patient will undergo preparation for surgery according to the standard care. Once anesthetized and intubated, electrodes will be attached to the patient's head. After placing the electrodes, when the patient is under anesthesia, a blood sample will be taken prior to BDF. This sample will be used as baseline for BDF. The patient will then undergo a BDF procedure. Additional blood samples will be taken post BDF for identification of CNS biomarkers. Surgery will then proceed according to the standard of care. Once the dura is opened, a CSF sample will be taken. The surgery will continue according to the standard of care. Adverse Events will be recorded according to CTCAE V 5.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects over the age of 18
* Able to sign informed consent
* Candidates for intradural tumor resection spinal surgery with intraoperative neuromonitoring.

Exclusion Criteria:

* Pacemakers, or other implanted electric medical devices
* Pregnant or lactating females
* Major medical, neurologic or psychiatric condition who are judged as unable to fully comply with the study
* History of skull fractures or previous brain surgery
* American Society of Anesthesiologists grade >2
* Anticoagulants treatment
* Damage to the dura resulting in CSF leak
* Patients with seizures/epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Elevation in blood concentration of CNS biomarkers following BDF compared to biomarkers detected in CSF of the same subject. The overall incidence of BDF procedure-related AEs and SAEs, with severity graded according to CTCAE v5.0 criteria. | Blood samples will be acquired before and 5 and 10 min post BDF. Another blood sample will be taken before opening the dura. CSF sample will be taken at the time of opening the dura.
  Efficacy We will quantify potential biomarkers in pre- and post- BDF blood samples and expect to see an increase in the blood concentration in the post-BDF samples. The primary endpoint of the study is the elevation in blood concentration of CNS biomarkers including fatty acid or other lipid levels, and/or barrier opening biomarkers and/or unique vascular and cytokines-related proteins and metabolites, following BDF, compared to biomarkers detected in cerebrospinal fluid (CSF) of the same subject.
  Safety The primary safety endpoint will be the overall incidence of BDF procedure-related AEs and SAEs, with severity graded according to CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ran Harel, MD, Principal Investigator — Sheba Medical Center; Yael Mardor, PhD, Study Chair — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in a published article (text, tables, figures, and appendices) will be available to qualified researchers upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal will receive the de-identified individual participant data that underlie the results reported in a published article (text, tables, figures, and appendices) by mail upon providing a methodologically sound proposal

REFERENCES:
- [Result] Sharabi S, Last D, Daniels D, Fabian ID, Atrakchi D, Bresler Y, Liraz-Zaltsman S, Cooper I, Mardor Y. Non-Invasive Low Pulsed Electrical Fields for Inducing BBB Disruption in Mice-Feasibility Demonstration. Pharmaceutics. 2021 Jan 27;13(2):169. doi: 10.3390/pharmaceutics13020169. PMID 33513968
- [Result] Sharabi S, Bresler Y, Ravid O, Shemesh C, Atrakchi D, Schnaider-Beeri M, Gosselet F, Dehouck L, Last D, Guez D, Daniels D, Mardor Y, Cooper I. Transient blood-brain barrier disruption is induced by low pulsed electrical fields in vitro: an analysis of permeability and trans-endothelial electric resistivity. Drug Deliv. 2019 Dec;26(1):459-469. doi: 10.1080/10717544.2019.1571123. PMID 30957567
- See also: Israeli ministry of health list of clinical trials — https://clinicaltrial.health.gov.il/clinicaltrials/?MOHResearchId=MOH_2025-08-11_014243